CLINICAL TRIAL: NCT01595269
Title: The Clinical and Economic Impacts of e-Heath on Diabetes
Acronym: eHealthDM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Danièle Pacaud (Individual)
Collaborators: The Lawson Foundation (Other)
Responsible Party: Sponsor-Investigator, Dr. Danièle Pacaud, Associate Professor, Pacaud, Danièle, M.D.
Organization: Pacaud, Danièle, M.D. (Individual)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: LAWSON-686
Record Dates: First submitted 2011-03-03; First posted 2012-05-10 (Estimated); Last update posted 2012-05-10 (Estimated); Status verified 2012-05

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Diabetes; eHealth; Type 2 Diabetes; Education; Calgary Health Region
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Education mode 1 (control) (Placebo Comparator): Education mode 1 (control) is comprised of participants educated using CHR's current traditional face-to-face delivery method, with printed materials and written log journals. These participants will be trained to use the University's web portal if they elect to access internet-based diabetes information. This allows for the tracking of the type and amounts of diabetes information accessed by participants.
  Interventions: Other: eHealth education
- Education mode 2 (static interface) (Active Comparator): Education mode 2 (static interface) participants will be educated using digitized forms of the traditional materials provided by CHR as well as an electronic log journal (e-journal) where participants will record their diabetes-related outcomes and behavioural information. Education mode 2 will be assessed and approved by CHR.
  Interventions: Other: eHealth education
- Education mode 3 (dynamic interface) (Active Comparator): Education mode 3 (dynamic interface) participants will be educated using the digitized traditional materials from education mode 2 as well as an enhanced dynamic e-journal (visualization of blood glucose and alerts). In addition, this mode will provide informative disease-related internet sites and diabetes news and articles vetted by the medical team. Participants and health professionals will then be able to electronically discuss the content and quality of this information (discussion board). New sites and articles will be added on an ongoing basis. Participants will also have access to a chat room that will encourage information sharing with other education mode 3 participants and health professionals at CHR. Education mode 3 will be assessed and approved by CHR.
  Interventions: Other: eHealth education

INTERVENTIONS:
Other: eHealth education — In addition to the face-to-face education process currently used at the CHR, Education mode 1 (control), Education mode 2 (static interface) and Education mode 3 (dynamic interface) will be used.

SUMMARY:
This project addresses the following Null Hypotheses:

1. There will be no difference will be found in the use of the search engine and the information accessed among the three education modes.
2. There will be no difference in education mode's effect on metabolic control, self-care management practices, and medical resource utilization.
3. There will be no difference in the economic impact on the health care system based on differing education modes.

DETAILED DESCRIPTION:
In addition to the face-to-face education process currently used at the CHR, this project will develop two modes of eHealth education. Education mode 1 (control) is comprised of participants educated using CHR's current traditional face-to-face delivery method, with printed materials and written log journals. These participants will be trained to use the University's web portal if they elect to access internet-based diabetes information. This allows for the tracking of the type and amounts of diabetes information accessed by participants. Education mode 2 (static interface) participants will be educated using digitized forms of the traditional materials provided by CHR as well as an electronic log journal (e-journal) where participants will record their diabetes-related outcomes and behavioural information. Education mode 2 will be assessed and approved by CHR. Education mode 3 (dynamic interface) participants will be educated using the digitized traditional materials from education mode 2 as well as an enhanced dynamic e-journal (visualization of blood glucose and alerts). In addition, this mode will provide informative disease-related internet sites and diabetes news and articles vetted by the medical team. Participants and health professionals will then be able to electronically discuss the content and quality of this information (discussion board). New sites and articles will be added on an ongoing basis. Participants will also have access to a chat room that will encourage information sharing with other education mode 3 participants and health professionals at CHR. Education mode 3 will be assessed and approved by CHR.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 or older
* Literate
* Not participating in other clinical trials
* Diabetes diagnosed within the last three months
* Type 2 diabetes
* No medical conditions that could compromise metabolic control
* No linguistic, cognitive or psychosocial barriers that would hinder study completion
* Computer and internet literate
* Access to high-speed internet

Exclusion Criteria:

* Under the age of 18
* Not literate
* Participating in other clinical trials
* Diabetes diagnosed greater than three months ago
* Type 1 diabetes
* Gestational diabetes
* Additional medical conditions that could compromise metabolic control
* Linguistic, cognitive or psychosocial barriers that would hinder study completion
* Not computer and internet literate
* No access to high-speed internet

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2007-04; Primary Completion 2008-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Changes in A1C | baseline, 3, 6, 9, 12 months
  A1C is a measure of metabolic control in diabetes. For this study changes in A1C from baseline to 3, 6, 9 and 12 months were measured. All A1C were measured in provincial laboratories using 6.1% as the upper limit of normal for individuals without diabetes.

SECONDARY OUTCOMES:
a reduction in the cost of delivering health information and education processes | baseline and 12 months
  Secondary effects could include a change in the cost of delivering health information and education processes. Potential changes to self-care management practices of people with type II diabetes could lead to a reduced utilization of the heath care system resulting in a positive economic impact.
Changes in Diabetes Knowledge | baseline, 3, 6, 9, 12 months
  Changes in diabetes knowledge from baseline to 3, 6, 9, and 12 months will be measured using a 23 item multiple choice questionnaire devolopped by Fitzgerald et al 1998.
Changes in Diabetes self-care activities | Baseline, 3, 6, 9 and 12 months
  Changes in diabetes self-care activities from base line to 3, 6, 9, and 12 months will be measured the diabetes self-care activities tool evaluated by Toobert at al (2000).

CONTACTS AND LOCATIONS:
Overall Officials: Angela M Downey, PhD, CMA, FCMA, Principal Investigator — University of Lethbridge; Helen Kelley, PhD, Principal Investigator — University of Lethbridge
Locations (1):
- Calgary Health Region's offices across southwestern Alberta, Lethbridge, Alberta, Canada